CLINICAL TRIAL: NCT03527264
Title: BrUOG 355: A Pilot Feasibility Study Incorporating Nivolumab to Tailored Radiation Therapy With Concomitant Cisplatin in the Treatment of Patients With Cervical Cancer
Brief Title: BrUOG 355: Nivolumab to Tailored Radiation Therapy With Concomitant Cisplatin in the Treatment of Patients With Cervical Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Brown University (Other)
Collaborators: Rhode Island Hospital (Other); The Miriam Hospital (Other); Women and Infants Hospital of Rhode Island (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 355
Record Dates: First submitted 2018-05-04; First posted 2018-05-17 (Actual); Results first posted 2022-04-26 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; Stage IB; Stage IIA; Stage IIB; Stage IIIA; Stage IIIB; Stage IVA
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Radiation; Nivolumab; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1A (Experimental): Nivolumab during Chemo/RT with whole pelvic RT
  Interventions: Drug: Nivolumab induction; Drug: Cisplatin; Radiation: Radiation; Drug: Nivolumab with chemoradiation
- Cohort 1B (Experimental): Nivolumab during Chemo/RT with extended field
  Interventions: Drug: Nivolumab induction; Drug: Cisplatin; Radiation: Radiation; Drug: Nivolumab with chemoradiation
- Cohort 2 (Experimental): Chemoradiation followed by Nivolumab Maintenance
  Interventions: Drug: Nivolumab induction; Drug: Cisplatin; Radiation: Radiation; Drug: Nivolumab maintenance
- Cohort 3 (Experimental): Nivolumab during chemoradiation and then as maintenance
  Interventions: Drug: Nivolumab induction; Drug: Cisplatin; Radiation: Radiation; Drug: Nivolumab with chemoradiation; Drug: Nivolumab maintenance

INTERVENTIONS:
Drug: Nivolumab induction — 2 doses Nivolumab 240mg IV
Drug: Cisplatin — 40 mg/m2 of cisplatin: Dosing on Days: 1, 8, 15, 22, 29, 36 beginning on day 1 of radiation therapy.
Radiation: Radiation — Total dose of 45 Gy in 25 fractions at 180 cGy/fx
  Whole pelvic or extended field
Drug: Nivolumab with chemoradiation — Nivolumab 240mg IV every 14 days (+/- 3 days) for 3 doses, administered concomitantly during chemoradiation and beginning day 1 of Radiation.
  Arms: Cohort 1A; Cohort 1B; Cohort 3
Drug: Nivolumab maintenance — Nivolumab 480 mg IV every 4 weeks for 2 years
  Arms: Cohort 2; Cohort 3

SUMMARY:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of the investigational drug in combination with radiation to learn whether the drug(s) works in treating a specific disease. In this study, researchers are studying three treatment arms, each using standard chemotherapy, with the drug cisplatin and radiation and the drug Nivolumab. Each treatment Arm will test the addition of Nivolumab at a different time point

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* ECOG performance status ≤2
* Patients with histologically confirmed advanced cervical cancer (any cell type): FIGO Clinical stages IB, IIA, IIB, IIIA, IIIB, IVA.
* Participants must have normal organ and marrow function as defined below:

  1. absolute neutrophil count ≥1,500/mcL
  2. platelets ≥100,000/mcL
  3. total bilirubin within normal institutional limits
  4. AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  5. creatinine Within normal institutional limits
* Neuropathy (sensory and motor) ≤ CTCAE v4.0 grade 1
* Patients with ureteral obstruction should undergo stent or nephrostomy tube placement prior to study entry. Any side effects or complications associated with stent placement that, in the opinion of the treating investigator, puts the patient at increased risk for treatment-related toxicity, must be resolved completely prior to study enrollment.
* Patients of child-bearing potential must have a negative serum pregnancy test prior to study entry (within 7 days prior to initiation of study treatment) and be practicing an effective form of contraception during study treatment and for 24 months (2 years) thereafter.
* Women should not breast-feed while on this study
* Patients must not be receiving any other investigational agent
* Ability to understand and the willingness to sign a written informed consent document.
* All patients with a history of hearing loss are required to have an audiogram within 28 days prior to initiating protocol therapy. If patient does not have a history of hearing loss this must be documented by treating physician.

Exclusion Criteria:

* Participants with visceral metastases, including brain metastases.
* Uncontrolled intercurrent illness
* Patients who have received previous pelvic or abdominal radiation, cytotoxic chemotherapy, or previous therapy of any kind for this malignancy
* Patients who have circumstances that will not permit completion of this study or the required follow-up as per the treating physician
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer are excluded if there is any evidence of other malignancy being present within the last three years (2 years for invasive breast cancer). However, patients with a malignancy that is non-likely to require treatment, as per the treating physician, in the next 2 years, such as a completely resected, early stage breast cancer, are eligible. Patients are also excluded if their previous cancer treatment contraindicates this protocol therapy.
* Prior treatment with immunotherapy for any cancer, including immune checkpoint inhibitors or anti-CTLA4 agents
* Patients with renal abnormalities, such as pelvic kidney, horseshoe kidney, or renal transplantation, that would require modification of radiation fields as documented by treating physician

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is for patients with cervical cancer, therefore all patients must be female
Enrollment: 4 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Don Dizon, MD, Principal Investigator — Brown University Oncology Research Group (BrUOG)
Locations (2):
- United States (2):
  - Rhode Island Hospital, Providence, Rhode Island
  - Women and Infants Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1A: Nivolumab during Chemo/RT with whole pelvic RT
  Nivolumab induction: 2 doses Nivolumab 240mg IV
  Cisplatin: 40 mg/m2 of cisplatin: Dosing on Days: 1, 8, 15, 22, 29, 36 beginning on day 1 of radiation therapy.
  Radiation: Total dose of 45 Gy in 25 fractions at 180 cGy/fx
  Whole pelvic or extended field
  Nivolumab with chemoradiation: Nivolumab 240mg IV every 14 days (+/- 3 days) for 3 doses, administered concomitantly during chemoradiation and beginning day 1 of Radiation.
- Cohort 1B: Nivolumab during Chemo/RT with extended field
  Nivolumab induction: 2 doses Nivolumab 240mg IV
  Cisplatin: 40 mg/m2 of cisplatin: Dosing on Days: 1, 8, 15, 22, 29, 36 beginning on day 1 of radiation therapy.
  Radiation: Total dose of 45 Gy in 25 fractions at 180 cGy/fx
  Whole pelvic or extended field
  Nivolumab with chemoradiation: Nivolumab 240mg IV every 14 days (+/- 3 days) for 3 doses, administered concomitantly during chemoradiation and beginning day 1 of Radiation.
- Cohort 2: Chemoradiation followed by Nivolumab Maintenance
  Nivolumab induction: 2 doses Nivolumab 240mg IV
  Cisplatin: 40 mg/m2 of cisplatin: Dosing on Days: 1, 8, 15, 22, 29, 36 beginning on day 1 of radiation therapy.
  Radiation: Total dose of 45 Gy in 25 fractions at 180 cGy/fx
  Whole pelvic or extended field
  Nivolumab maintenance: Nivolumab 480 mg IV every 4 weeks for 2 years
- Cohort 3: Nivolumab during chemoradiation and then as maintenance
  Nivolumab induction: 2 doses Nivolumab 240mg IV
  Cisplatin: 40 mg/m2 of cisplatin: Dosing on Days: 1, 8, 15, 22, 29, 36 beginning on day 1 of radiation therapy.
  Radiation: Total dose of 45 Gy in 25 fractions at 180 cGy/fx
  Whole pelvic or extended field
  Nivolumab with chemoradiation: Nivolumab 240mg IV every 14 days (+/- 3 days) for 3 doses, administered concomitantly during chemoradiation and beginning day 1 of Radiation.
  Nivolumab maintenance: Nivolumab 480 mg IV every 4 weeks for 2 years
Period: Overall Study
Arm/Group | Cohort 1A | Cohort 1B | Cohort 2 | Cohort 3
Started | 3 | 1 | 0 | 0
Completed | 3 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was terminated prior to enrolling patients in cohort 2 & cohort 3.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1A | Cohort 1B | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 3 | 1 | 0 | 0 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  |  | 0
  Between 18 and 65 years | 1 | 1 |  |  | 2
  >=65 years | 2 | 0 |  |  | 2
Age, Continuous [Mean (Full Range); unit: years] | 66 [62 to 69] | 54 [54 to 54] |  |  | 63 [54 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 |  |  | 4
  Male | 0 | 0 |  |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 |  |  | 1
  Not Hispanic or Latino | 2 | 1 |  |  | 3
  Unknown or Not Reported | 0 | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  |  | 0
  Asian | 0 | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
  Black or African American | 0 | 0 |  |  | 0
  White | 2 | 1 |  |  | 3
  More than one race | 0 | 0 |  |  | 0
  Unknown or Not Reported | 1 | 0 |  |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 |  |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Number of patients that are alive without disease progression at time of analysis.
Time Frame: From start of study treatment through date of study completion, an average of 2 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A | Cohort 1B
Number analyzed (Participants) | 3 | 1
Participants | 2 | 1

2. Secondary Outcome: Recurrence Patterns
Description: Determination of the site of recurrence, loco-regional versus distant
Time Frame: From start of study treatment through date of study completion, an average of 2 years.
Population: Only 1 patient on cohort 1A had recurrence within 3 years of study entry.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A | Cohort 1B
Number analyzed (Participants) | 1 | 0
Participants
  Loco-regional | 1 | 0
  Distant | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events were reported from the time a signed and dated ICF is obtained through study treatment completion, an average of 6 months.
Arm/Group | Cohort 1A | Cohort 1B
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/1
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1A (N=3) | Cohort 1B (N=1)
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Generalized muscle weakness (General disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1A (N=3) | Cohort 1B (N=1)
Anemia (Blood and lymphatic system disorders) | 3 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Dizziness (Psychiatric disorders) | 1 | 1
Weight loss (Investigations) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Lipase increased (Investigations) | 1 | 1
Lymphocyte count decreased (Investigations) | 3 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0
White blood cell count decreased (Investigations) | 3 | 0
Neutrophil count decreased (Investigations) | 2 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Hypoalbuminemia (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 2 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
GERD (Gastrointestinal disorders) | 1 | 0
Serum amylase increased (Investigations) | 1 | 0
Serum creatinine increased (Investigations) | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Cough (General disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypocalcemia (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT03527264/Prot_SAP_ICF_000.pdf